CLINICAL TRIAL: NCT04294940
Title: Impact of a Digital Solution (CardiCare™) on Cardiorespiratory Fitness Improvement in Patients Discharged From a Phase 2 Cardiac Rehabilitation Following an Acute Coronary Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to the COVID-19 pandemic. Some study procedures are not curently possible for many investigational sites.
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CardiCare
Record Dates: First submitted 2020-02-25; First posted 2020-03-04 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Acute Coronary Syndrome
Keywords: CardiCare; Coronary heart disease; Application; Mobile; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: standard of care (Other): The patient will follow the hygiene-dietetic recommendations given by their centre and wear an actigraph night and day.
  Interventions: Other: Wear an actigraph
- Group B: standard of care + mobile application CardiCare™ (Other): The patient will follow the hygiene-dietetic recommendations given by their centre, wear an actigraph night and day and use the mobile application CardiCare™
  Interventions: Other: Use the mobile application CardiCare™ and wear an actigraph

INTERVENTIONS:
Other: Wear an actigraph — Between visits, tha patient will have to:
  * Follow the hygiene-dietetic recommendations given by their centre.
  * Wear the actigraph night and day Patients
  Arms: Group A: standard of care
Other: Use the mobile application CardiCare™ and wear an actigraph — Between visits, tha patient will have to:
  * Follow the hygiene-dietetic recommendations given by their centre.
  * Wear the actigraph night and day Patients
  * wear their smartphone everyday and use the mobile application CardiCare™
  Arms: Group B: standard of care + mobile application CardiCare™

SUMMARY:
Coronary heart disease is a partial inability of the coronary arteries to supply the heart muscle due to their narrowing. There is angina and myocardial infarction. Coronary heart disease is the first cause of non-communicated deaths and years of life lost.

After hospital discharge, a few days following the acute care of a coronary heart disease, a formal Cardiac Rehabilitation programme (CR) is usually provided. CR is a comprehensive programme involving exercise training, risk factor modification, education and psychological support. It is generally sequenced in 4 phases. Phase 1 begins at the hospital and consists of early mobilisation and education. Most phase 2 CR models are based upon supervised ambulatory outpatient programmes. Maintenance (phase 3 and 4) follows the ambulatory programme in which physical fitness and risk factor control are supported in a minimally supervised setting.

Despite high-grade recommendations and abundant clinical evidence, a CR program is not always implemented and the patients are not systematically referred after discharge from a phase 1 CR. Furthermore, compliance to pharmacological treatments and changes in lifestyle and diet are hugely neglected following a phase 2 CR and an important number of patients resume a sedentary lifestyle.

A growing body of evidence supports the use of digital tools such as smartphones and tablets in helping the patients achieve their goals in terms of physical exercise, risk-factor reduction and diet improvement.

Ad Scientiam has developed CardiCare™, a mobile application intended to provide a personalised physical training plan contributing to stabilise or improve cardiorespiratory fitness through improvement of VO2max.

The mobile application CardiCare™ is to be used by patients after an acute coronary syndrome, graduated from a phase 2 cardiac rehabilitation program in a cardiac rehabilitation centre and entering in phase 3 CR.

The mobile application CardiCare™ consists of several modules:

* A physical activity recommendation engine, providing personalised weekly activity schedule, self-adapting to the patient's clinical characteristics, physical capacity and sport preferences through a proprietary algorithm
* Self-administered questionnaires to assess perceived exertion, chest pain, weight variations, patient's quality of life
* Passive monitoring of the patient's physical activity through Apple's HealthKit and Google's Fit
* Informational content about cardiovascular diseases, risk factor reduction and chest pain action plan The investigator's work hypothesis is that, compared to standard care, CardiCare™ will stabilise or improve the cardiorespiratory fitness (VO2max) acquired post-CR.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years old.
* Diagnosis of an Acute Coronary Syndrome in the last 3 months, documented by angiographically-proven coronary artery disease or hospitalisation report.
* Graduated from a phase 2 cardiac rehabilitation, ready to enter a phase 3 CR at home.
* Having agreed to perform a cardiopulmonary exercise testing and blood count at the inclusion or having performed a cardiopulmonary exercise testing and blood count within the last week.
* Owning a personal smartphone (Android 5.0 or beyond / iPhone 5s and newer supporting IOS 12 and beyond) with Wifi or a data plan (3G/4G).
* Able to use a smartphone (e.g. no vision, hearing, cognitive or dexterity impairment).
* Having agreed to install CardiCare™ application on their own smartphone.
* Having agreed to wear an actigraph at all times and install the actigraph application (CenterPoint Sync) on their smartphone.
* Enrolled in or benefiting of a national health system.
* Having read the information sheet and signed the informed consent form.

Non-inclusion Criteria:

* Treated with Coronary Artery Bypass Grafting.
* Cardiac surgery in the last 12 weeks.
* Planned revascularisation or surgery in the next 6 months.
* Clinical heart failure or Left Ventricular Ejection Fraction < 40% documented within the last 2 months.
* Severe valvular disease.
* Severe pulmonary disease.
* Chronic kidney disease (stages III-V).
* Drug or/and alcohol abuse (as per clinician's judgment).
* Unstable angina.
* Osteoarticular condition or other reasons that limit exercise for more than 4 months (clinician's judgment).
* Uncontrolled hypertension (resting Diastolic BP>100 mmHg and resting Systolic BP >200 mmHg).
* Severe/uncontrolled arrhythmia.
* Systemic medical diseases that are likely to affect cognitive functioning.
* Pregnant women confirmed by a pregnancy test at the inclusion.
* Participation to another interventional clinical trial (category 1).
* Illiterate or not proficient in the language of the study country (French, Italian, Spanish or Portuguese according to the country).
* Person under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy at 6 months of CardiCare™ in stabilising or improving the Cardiorespiratory Fitness of patients after acute coronary syndrome, graduated from a phase 2 cardiac rehabilitation program, versus standard care. | From day 0 to month 6
  Proportion of participants with stabilised or improved VO2max 6 months, as measured by Cardiopulmonary Exercise Test in group B versus group A

SECONDARY OUTCOMES:
To evaluate CardiCare™ impact on global physical activity between both groups over time of follow-up. | From day 0 to month 6
  The global physical activity will be monitored using continuous variables of the actigraph
To evaluate CardiCare™ impact on change in cardiorespiratory fitness at 3 months versus baseline in both groups. | From day 0 to month 3
  Proportion of participants in group B versus group A with stabilised or improved VO2max at 3 months compared to baseline.
To evaluate CardiCare™ impact on change in other cardiorespiratory fitness parameters at 3 and 6 months versus baseline, in both groups | From day 0 to month 3 and month 6
  Comparison in continous measurement of cardiorespiratory fitness as measured by Cardiopulmonary Exercise Test
To evaluate CardiCare™ impact on change in lipid levels at 3 and 6 months versus baseline, in both groups. | From day 0 to month 3 and month 6
  Identification of items will be based in continuous measurement of total cholesterol, Low Density Lipoproteins Cholesterol, High Density lipoproteins Cholesterol.
To evaluate CardiCare™ impact on change in glucose levels at 3 and 6 months versus baseline, in both groups. | From day 0 to month 3 and month 6
  Identification of items will be based in continuous measurement of fasting glucose
To evaluate CardiCare™ impact on change in weight at 3 months and 6 months versus baseline in both groups. | From day 0 to month 3 and month 6
  Identification of items will be based on measured clinical exam
To evaluate CardiCare™ impact on change in Body Mass Index at 3 months and 6 months versus baseline in both groups. | From day 0 to month 3 and month 6
  Identification of items will be based on measured clinical exam
To evaluate CardiCare™ impact on change in Hip and waist circumference at 3 months and 6 months versus baseline in both groups. | From day 0 to month 3 and month 6
  Identification of items will be based on measured clinical exam
To evaluate the impact of CardiCare™ on anxiety at 3 and 6 months versus baseline, in both groups. | From day 0 to month 3 and month 6
  Identification of the items will be measure with Hospital Anxiety and Depression Scale questionnaires
To evaluate the impact of CardiCare™ on quality of life at 3 and 6 months versus baseline, in both groups. | From day 0 to month 3 and month 6
  Identification of the items will be measure with Health-Related Quality of Life questionnaires
To evaluate medication compliance in both groups. | From day 0 to month 6
  Compliance will based on the duration of medication interruption.
To compare differences of reported cardiovascular events at 3 and 6 months, in both groups. | From day 0 to month 3 and month 6
  Comparison will based on the number of cardiovascular events occured
To compare time to first hospital readmission among both groups (all-cause, cardiac, and noncardiac) and their predictors. | From day 0 to month 3 and month 6
  Comparison will based on the number of hospital readmission
To assess the cost-effectiveness to reduce 30-day, 3 months and 6 months readmission rates using CardiCare™ as an intervention compared to standard care. | From day 0 to month 3 and month 6
  Identification of the items based on the number of hospital readmission
To evaluate the impact of CardiCare™ on employment status at 3 and 6 months versus baseline in both groups. | From day 0 to month 3 and month 6
  Identification of the items will based on the time to return to work and the time in sick leave
To evaluate CardiCare™ impact on exercise performed in group B. | From day 0 to month 6
  Comparison of the exercise performed during the follow up of participants in group B.
To evaluate CardiCare™ impact on cardiovascular risk factors control at 3 and 6 months versus baseline in both groups. | From day 0 to month 3 and month 6
  Identification of the cardiovascular risk factors will based on the clinical exam and blood tests
To evaluate, for each session, the correlation between self-reported physical activities in CardiCare™ and those collected by the actigraph in group B. | From day 0 to month 6
  Identification of items will be based on the physical activities reported by the patient in CardiCare™ and actigraph
To identify patterns of VO2max evolution between D0, M3 and M6, between both groups | From day 0 to month 3 and month 6
  Identification of items will be based on the measures of cardiorespiratory fitness as measured by Cardiopulmonary Exercise Test
To evaluate CardiCare™ impact on sleep quality between groups over time of follow-up. | From day 0 to month 6
  Identification of the items be based on actigraph
To evaluate the safety of the CardiCare™ use. | From day 0 to month 6
  Safety will be assessed by the numbers of adverse events and adverse events related to the use of the application CardiCare™.
To collect patients and investigators feedback on the CardiCare™ application. | From day 0 to month 6
  Descriptive analysis of patients and investigators satisfaction related to the mobile application.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Cohen Solal, Prof, Principal Investigator — Lariboisière Hospital
Locations (10):
- France (4):
  - Corentin Celton hospital, Issy-les-Moulineaux
  - Lariboisière hospital, Paris
  - Saint-Yves clinic, Rennes
  - Brie Cardiac Readaptation Centre, Villeneuve-Saint-Denis
- Italy (2):
  - Maugeri Scientific Clinical Institutes, Pavia
  - Scientific Institute of Hospitalization and Care San Raffaele Pisana, Roma
- Portugal (2):
  - CHOL - Santa Cruz hospital, Carnaxide
  - CHULN - Santa Marta hospital, Lisbon
- Spain (2):
  - Carlos III - La Paz Hospital, Madrid
  - Santiago University Hospital, Santiago de Compostela

REFERENCES:
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536